CLINICAL TRIAL: NCT00097227
Title: A Randomized Phase II Trial of Two Dose Schedules of Carboplatin/Paclitaxel/Cetuximab in Stage IIIB/IV Non-small Cell Lung Cancer
Brief Title: Trial of Carboplatin/Paclitaxel/Cetuximab in Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA225-058
Record Dates: First submitted 2004-11-18; First posted 2004-11-19 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; non-small; lung; IIIb; IV; Carboplatin; Paclitaxel; Cetuximab; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (3-week cycle) (Active Comparator): Cetuximab was administered weekly at an initial dose (Week 1) of 400 mg/m2 IV infusion and a weekly maintenance dose of 250 mg/m2 IV infusion.
  Paclitaxel 225 mg/m2 infused over 180 minutes on Day 1 and subsequently every 3 weeks.
  Carboplatin (AUC = 6) was infused over 30 minutes on Day 1 and subsequently every 3 weeks.
  Interventions: Biological: Cetuximab; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (4-week cycle) (Active Comparator): Cetuximab was administered weekly at an initial dose (Week 1) of 400 mg/m2 IV infusion and a weekly maintenance dose of 250 mg/m2 IV infusion.
  Paclitaxel 100 mg/m2 infused over 180 minutes on Day 1, Day 8 and Day 15 of a 4-week cycle.
  Carboplatin (AUC = 6) was infused over 30 minutes on Day 1 and subsequently every 4 weeks.
  Interventions: Biological: Cetuximab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Cetuximab — (Week 1) of 400 mg/m2 IV infusion and a weekly maintenance dose of 250 mg/m2 IV infusion.
  A cycle of therapy was defined as 3 weeks in Arm A and 4 weeks in Arm B.
  Other Names: Erbitux
Drug: Carboplatin — (AUC = 6) was infused over 30 minutes on Day 1 and subsequently every 3 weeks (AUC = 6) was infused over 30 minutes on Day 1 and subsequently every 4 weeks.
  Other Names: Paraplatin
Drug: Paclitaxel — 225 mg/m2 infused over 180 minutes on Day 1 and subsequently every 3 weeks. OR 100 mg/m2 infused over 180 minutes on Day 1, Day 8 and Day 15 of a 4-week cycle.
  Other Names: Taxol

SUMMARY:
The purpose of the study is to determine if the combination of cetuximab, carboplatin and paclitaxel will shrink a specific type of lung cancer known as non-small cell lung cancer (NSCLC). The safety of this combination will also be evaluated.

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer diagnosed for both genders in the United States. Approximately 173,770 new cases are estimated for 2004. It is the leading cause of cancer deaths in both men and women, with approximately 160,440 deaths estimated for 2004. Prognosis for many is poor if not diagnosed at an early stage, and therapy for advanced disease is limited. The study will test two chemotherapy agents, carboplatin and paclitaxel, in combination with a newly approved drug called cetuximab, which is continuing to be tested in colorectal cancer and other cancers. Cetuximab is a monoclonal antibody, which is believed to work by attaching to an epidermal growth factor receptor (EGFR) on tumor cells and thereby blocking tumor cells from reproducing. It is an antibody to the EGFR. Fifty percent of lung cancers overexpress EGFR.

Rationale:

The present study is built upon the data from previous studies, incorporating cetuximab into each of two regimens of paclitaxel plus carboplatin. The results of prior studies using paclitaxel and carboplatin demonstrate that these drugs in combination, using a variety of schedules, are both safe and effective as therapy for advanced or metastatic NSCLC. The addition of biologic therapy with the anti-EGFR agent cetuximab to the combination will presumably maximize the therapeutic index while keeping toxicity to a minimum in patients with Stage IIIB/IV NSCLC.

Research Hypothesis:

Subjects with previously-untreated stage IIIB/IV NSCLC who receive a combination of paclitaxel, carboplatin, and cetuximab will have a progression-free survival rate greater than that previously reported for subjects receiving the combination of paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects must fulfill all of the following criteria and have a complete signed informed consent form.

* Subjects must have signed an approved informed consent.
* Subjects with histologically or cytologically documented stage IIIB (supraclavicular lymph node, high neck node, or pleural effusion involvement) or IV NSCLC. Disease must be newly diagnosed or recurrent at least 1 year post adjuvant therapy.
* Subjects with measurable disease.
* Subjects with ECOG performance status 0-1.
* Subjects with asymptomatic brain metastasis are eligible; however, they must have completed radiotherapy/radiosurgery at least 2 weeks prior to enrollment and be off steroids.
* Radiotherapy must have been completed > 2 weeks prior to enrollment and the subject must have recovered from all adverse effects of prior radiotherapy. No previous irradiation to the only area of measurable disease. New lesions that developed in a previously irradiated area will be allowed.
* If diagnostic tissue or slides are available for a subject, these must be submitted for testing of EGFR status.
* Subjects ≥18 years of age.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level >35mIU/mL]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.
* Subjects with adequate hematologic function defined as: ANC ≥1,500/mm 3 ; WBC

  ≥3,000/mm 3 ; platelets ≥100,000/mm 3 ; and hemoglobin ≥9 g/dL.
* Subjects with adequate hepatic function defined as: total bilirubin ≤1.5 x upper limit of normal (ULN) or AST ≤2.5 x ULN.
* Subjects with adequate renal function defined as a serum creatinine level ≤1.5 mg/dL or a creatinine clearance ≥60 cc/minute.

Exclusion Criteria:

Any of the following criteria will make the subject ineligible to participate in this study.

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study. Subjects who are men must also agree to use effective contraception.
* WOCBP using a prohibited contraceptive method.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Subjects who have had prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 years.
* Subjects with significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure, cardiomyopathy with decreased ejection fraction, myocardial infarction within the past year, or cardiac ventricular arrythmias requiring medication.
* Subjects with an uncontrolled seizure disorder, or active neurological disease.
* Subjects with symptomatic brain metastasis. Prohibited Therapies and/or Medications
* Subjects who have received prior systemic chemotherapy. Subjects with no more than one prior adjuvant regimen for initially diagnosed disease are eligible for the study.
* Subjects with a history of prior cetuximab or other therapy that specifically and directly targets the EGFR pathway.
* Subject with prior severe infusion reaction to a monoclonal antibody.
* Subjects with know allergy to Cremophor EL.
* Subjects with known peripheral neuropathy (> grade 1).
* Subjects with prior erythropoietin (i.e., Epogen, Procrit) treatment.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To estimate median progression free survival and the progression free survival rate | 6 months

SECONDARY OUTCOMES:
To estimate the overall response rate in each treatment arm | 6 months
To estimate median survival and the survival rate at one year in each treatment arm | 6 months
To evaluate the toxicity profile of each treatment arm | 6 months
To explore the relationship between EGFR expression and the "clinical benefit" received from each treatment regimen | 6 months
To evaluate symptom response rate in each treatment arm using the Lung Cancer Subscale (LCS) of the FACT-L | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (20):
- United States (20):
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Santa Monica, California
  - ImClone Investigational Site, Newark, Delaware
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, St. Petersburg, Florida
  - ImClone Investigational Site, Tucker, Georgia
  - ImClone Investigational Site, Terra Haute, Indiana
  - ImClone Investigational Site, Louisville, Kentucky
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Ypsilanti, Michigan
  - ImClone Investigational Site, Newark, New Jersey
  - ImClone Investigational Site, Chapel Hill, North Carolina
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Columbia, South Carolina
  - ImClone Investigational Site, Knoxville, Tennessee
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Temple, Texas
  - ImClone Investigational Site, Richmond, Virginia
  - ImClone Investigational Site, Tacoma, Washington
  - ImClone Investigational Site, Morgantown, West Virginia